CLINICAL TRIAL: NCT02717806
Title: Technology-enabled Cardiac Rehabilitation Through PATHway. Feasibility, Clinical Effectiveness and Cost-effectiveness
Acronym: PATHway
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Collaborators: Dublin City University (Other)
Responsible Party: Principal Investigator, Roselien Buys, Dr, KU Leuven
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: S59023
Record Dates: First submitted 2016-03-18; First posted 2016-03-24 (Estimated); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Cardiovascular Disease
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PATHway (Experimental): Patients allocated to the PATHway intervention will be given a 4 week run-in period as an outpatient to get acquainted with the system. During this run-in period, the PATHway system will also be installed in each participant's home. They will be provided with a training manual and a quick set up guide for getting started with PATHway in the home.
  After this 4 week run-in period, the PATHway system will be set up for each individual patient including a patient specific exercise prescription. The patient will then exercise with the PATHway platform for 6 months.
  Interventions: Behavioral: PATHway
- Usual care (No Intervention): Patients randomized to the control group will receive usual care.

INTERVENTIONS:
Behavioral: PATHway — Patients will use the PATHway platform for 6 months
  Arms: PATHway

SUMMARY:
The PATHway system is designed to help patients remain physically active and maintain a good cardiovascular health. It proposes a novel approach that aims to empower patients to self-manage their CVD, set within a collaborative care context with health professionals. This will be achieved via a patient-centric holistic approach that specifically addresses the above barriers. It involves an internet-enabled and sensor-based home exercise platform. It is represented by several modules with an exercise module as the core component which will provide individualized rehabilitation programs that use regular, socially inclusive exercise sessions as the basis upon which to provide a personalized, comprehensive lifestyle intervention program (managing exercise, smoking, diet, stress, alcohol use etc.) to enable patients to both better understand and deal with their own condition and to lead a healthier lifestyle in general.

The goal of this trial is to assess the acceptability, short-term effectiveness on lifestyle and health related physical fitness and cost-effectiveness of the PATHway intervention in patients with CVD in a single blind multicentre pilot randomised controlled trial (RCT).

ELIGIBILITY:
Inclusion Criteria:

* Men and women with documented CVD
* age 40-80 yrs
* patients are on optimal medical treatment and stable with regard to symptoms and pharmacotherapy for at least 4 weeks
* patients must have completed the ambulatory CR program and received clinical approval from their treating physician to continue exercising outside the hospital program
* internet access at home

Exclusion Criteria:

* significant illness during the last 6 weeks
* known severe ventricular arrhythmia with functional or prognostic significance
* significant myocardial ischemia, hemodynamic deterioration or exercise-induced arrhythmia at baseline testing
* cardiac disease that limits exercise tolerance (valve disease with significant hemodynamic consequences, hypertrophic cardiomyopathy etc.)
* co-morbidity that may significantly influence one-year prognosis
* functional or mental disability that may limit exercise
* acute or chronic inflammatory diseases or malignancy, the use of anti-inflammatory drugs or immune suppression
* GFR <25ml/min/1.73m2
* hemoglobin < 10g/dl
* severe chronic obstructive pulmonary disease (FEV1 < 50%)
* NYHA class 4
* participation in another clinical trial

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Change in total volume of weekly active energy expenditure | 3 and 6 months

CONTACTS AND LOCATIONS:
Locations (3):
- University Hospitals Leuven, Leuven, Belgium
- Ireland (2):
  - Beaumont Hospital, Dublin
  - Mater Misericordiae Hospital, Dublin

REFERENCES:
- [Derived] Claes J, Cornelissen V, McDermott C, Moyna N, Pattyn N, Cornelis N, Gallagher A, McCormack C, Newton H, Gillain A, Budts W, Goetschalckx K, Woods C, Moran K, Buys R. Feasibility, Acceptability, and Clinical Effectiveness of a Technology-Enabled Cardiac Rehabilitation Platform (Physical Activity Toward Health-I): Randomized Controlled Trial. J Med Internet Res. 2020 Feb 4;22(2):e14221. doi: 10.2196/14221. PMID 32014842
- [Derived] Claes J, Buys R, Woods C, Briggs A, Geue C, Aitken M, Moyna N, Moran K, McCaffrey N, Chouvarda I, Walsh D, Budts W, Filos D, Triantafyllidis A, Maglaveras N, Cornelissen VA. PATHway I: design and rationale for the investigation of the feasibility, clinical effectiveness and cost-effectiveness of a technology-enabled cardiac rehabilitation platform. BMJ Open. 2017 Jun 30;7(6):e016781. doi: 10.1136/bmjopen-2017-016781. PMID 28667228